CLINICAL TRIAL: NCT01940900
Title: A Phase 3 Randomized, Double-masked, Controlled Trial to Establish the Safety and Efficacy of Intravitreous Administration of Fovista® (Anti PDGF-B Pegylated Aptamer) Administered in Combination With Lucentis® Compared to Lucentis® Monotherapy in Subjects With Subfoveal Neovascular Age-related Macular Degeneration.
Brief Title: A Phase 3 Safety and Efficacy Study of Fovista® (E10030) Intravitreous Administration in Combination With Lucentis® Compared to Lucentis® Monotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPH1003
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2018-08

CONDITIONS: Age-Related Macular Degeneration
Keywords: Wet AMD; choroidal neovascularization; Fovista®; E10030; Lucentis®
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — E10030 aptamer; Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E10030 + ranibizumab (Experimental): E10030 1.5 mg intravitreal injection + ranibizumab 0.5 mg intravitreal injection
  Interventions: Drug: E10030; Drug: ranibizumab
- Sham + ranibizumab (Active Comparator): E10030 sham intravitreal injection + ranibizumab 0.5 mg intravitreal injection
  Interventions: Drug: ranibizumab; Drug: E10030 sham intravitreal injection

INTERVENTIONS:
Drug: E10030
  Other Names: Fovista®
  Arms: E10030 + ranibizumab
Drug: ranibizumab
  Other Names: Lucentis®
Drug: E10030 sham intravitreal injection — Pressure on the eye with a syringe with no needle
  Other Names: Sham
  Arms: Sham + ranibizumab

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of intravitreal administration of Fovista® administered in combination with Lucentis® compared to Lucentis® monotherapy in subjects with subfoveal choroidal neovascularization secondary to age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio to the following dose groups:

* Fovista® 1.5 mg/eye + Lucentis® 0.5 mg/eye
* Fovista® sham + Lucentis® 0.5 mg/eye

Subjects will be treated for a total of 24 months with active Fovista® or sham in combination with Lucentis® with the primary endpoint at 12 months.

Primary Efficacy Endpoint:

The primary efficacy endpoint is the mean change in visual acuity (ETDRS letters) from baseline at the month 12 visit.

Safety Endpoints:

Safety endpoints include adverse events, vital signs, ophthalmic variables [ophthalmic examination, intraocular pressure (IOP), fluorescein angiogram (FA), optical coherence tomography (OCT)], ECG, and laboratory variables.

Approximately 622 subjects will be randomized into one of the two treatment cohorts (311 patients per dose group).

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender aged ≥ 50 years
* Active subfoveal choroidal neovascularization (CNV) secondary to AMD
* Presence of sub-retinal hyper-reflective material (SD-OCT)

Exclusion Criteria:

* Any prior treatment for AMD in the study eye prior to the Day 1 visit, except oral supplements of vitamins and minerals
* Any prior intravitreal treatment in the study eye prior to the Day 1 visit, regardless of indication (including intravitreal corticosteroids)
* Any intraocular surgery or thermal laser within three (3) months of trial entry. Any prior thermal laser in the macular region, regardless of indication
* Subjects with subfoveal scar or subfoveal atrophy are excluded
* Diabetes mellitus

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (104):
- United States (46):
  - Tucson, Arizona
  - Fresno, California
  - La Jolla, California
  - Loma Linda, California
  - Mountain View, California
  - Sacramento, California
  - Santa Ana, California
  - Aurora, Colorado
  - Golden, Colorado
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Largo, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Harvey, Illinois
  - West Des Moines, Iowa
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Peabody, Massachusetts
  - Worcester, Massachusetts
  - Minneapolis, Minnesota
  - Lawrenceville, New Jersey
  - New York, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Greenville, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Bellevue, Washington
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Santa Fe
- Australia (6):
  - East Melbourne
  - Malvern
  - Nedlands
  - Parramatta
  - Sydney
  - Westmead
- Colombia (3):
  - Bogotá
  - Cali
  - Medellín
- Denmark (5):
  - Aalborg
  - Aarhus C
  - Glostrup Municipality
  - Odense
  - Roskilde
- France (7):
  - Créteil
  - Lyon
  - Marseille
  - Paris
  - Rouen
  - Strasbourg
  - Tours
- Germany (15):
  - Aachen
  - Bonn
  - Cologne
  - Freiburg im Breisgau
  - Göttingen
  - Hamburg
  - Heidelberg
  - Karlsruhe
  - Kiel
  - Leipzig
  - Lübeck
  - Mainz
  - München
  - Münster
  - Tübingen
- Hungary (5):
  - Budapest
  - Debrecen
  - Magyarszék
  - Pécs
  - Szeged
- Israel (6):
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Rehovot
  - Tel Aviv
- Spain (6):
  - Barcelona
  - Bilbao
  - Las Palmas
  - Navarro
  - Sant Cugat del Vallès
  - Valencia
- Turkey (Türkiye) (2):
  - Ankara
  - Izmir

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 627 patients were randomized but 1 patient was not treated
Groups:
- E10030 + Ranibizumab: E10030 1.5 mg intravitreal injection + ranibizumab 0.5 mg intravitreal injection
  E10030
  ranibizumab
- Sham + Ranibizumab: E10030 sham intravitreal injection + ranibizumab 0.5 mg intravitreal injection
  ranibizumab
  E10030 sham intravitreal injection: Pressure on the eye with a syringe with no needle
Period: Overall Study
Arm/Group | E10030 + Ranibizumab | Sham + Ranibizumab
Started | 311 | 315
Completed | 282 | 284
Not Completed | 29 | 31
Not completed — Physician Decision | 4 | 0
Not completed — Adverse Event | 10 | 15
Not completed — Withdrawal by Subject | 11 | 15
Not completed — Lost to Follow-up | 1 | 0
Not completed — Sponsor Decision | 1 | 0
Not completed — subject non-compliance | 1 | 1
Not completed — other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E10030 + Ranibizumab | Sham + Ranibizumab | Total
Number analyzed (Participants) | 311 | 315 | 626
Age, Customized [Count of Participants; unit: Participants]
  Age: Adults 18-64 years | 30 | 31 | 61
  Age: Adults 65-84 years | 224 | 221 | 445
  Age: Adults 85 years and over | 57 | 63 | 120
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 189 | 367
  Male | 133 | 126 | 259
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 11 | 9 | 20
  Argentina | 21 | 15 | 36
  Turkey | 3 | 4 | 7
  Hungary | 58 | 61 | 119
  United States | 100 | 97 | 197
  Denmark | 11 | 12 | 23
  Israel | 34 | 31 | 65
  Australia | 4 | 9 | 13
  France | 49 | 55 | 104
  Germany | 8 | 9 | 17
  Spain | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity From Baseline to 12 Months
Description: The primary efficacy endpoint is the mean change in visual acuity (ETDRS letters) from baseline to the month 12 visit. Higher ETDRS letters represents higher vision and a higher change in ETDRS letters represents better functioning.
Time Frame: 12 Months
Population: Mean change in visual acuity (ETDRS letter) from Baseline to Month 12
Measure: Mean (Standard Error); unit: letters
Arm/Group | E10030 + Ranibizumab | Sham + Ranibizumab
Number analyzed (Participants) | 311 | 315
letters | 9.91 (0.88) | 10.36 (0.87)

ADVERSE EVENTS:
Time Frame: Up to 12 months of exposure
Description: The efficacy (ITT) population, defined as all subjects randomized and received at least one dose of study drug, is different than the safety population, where all subjects who have received at least one dose of E10030 are analyzed as on that group. There was one subject who was randomized to Sham+Ranibizumab but was mis-treated with one dose of E10030 and therefore was analyzed in the E10030+ranibizuma group for safety purposes. This is the same explanation for the SAE and Mortality tables.
Arm/Group | E10030 + Ranibizumab | Sham + Ranibizumab
All-Cause Mortality (participants affected / at risk) | 4/312 | 4/314
Serious Adverse Events (participants affected / at risk) | 56/312 | 49/314
Other Adverse Events (participants affected / at risk) | 161/312 | 136/314
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E10030 + Ranibizumab (N=312) | Sham + Ranibizumab (N=314)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Follicle centre, lymphoma, follicular grade I, II, III stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 3 (3)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (3) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cataract traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (4)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Macular hole (Eye disorders) | 3 (3) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 3 (4) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Retinal pigment epithelial tear (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Chlostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 6 (6) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E10030 + Ranibizumab (N=312) | Sham + Ranibizumab (N=314)
Conjunctival haemorrhage (Eye disorders) | 74 (166) | 50 (136)
Punctate keratitis (Eye disorders) | 35 (93) | 40 (97)
Conjuctival hyperaemia (Eye disorders) | 24 (48) | 24 (53)
Eye pain (Eye disorders) | 22 (51) | 21 (35)
Vitreous floaters (Eye disorders) | 22 (28) | 12 (13)
Eye irritation (Eye disorders) | 18 (34) | 15 (35)
Keratitis (Eye disorders) | 18 (64) | 14 (47)
Nasopharyngitis (Infections and infestations) | 17 (18) | 18 (20)
Urinary tract infection (Infections and infestations) | 17 (23) | 18 (25)
Bronchitis (Infections and infestations) | 16 (18) | 11 (12)
Intraocular pressure increased (Investigations) | 49 (101) | 25 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution agrees not to individually publish the results of the Study without Ophthotech's prior written consent. Institution may participate in a joint, multi-center publication of the Study results with other investigators and/or institutions only, upon the prior written consent of Ophthotech.